CLINICAL TRIAL: NCT05690815
Title: Express Testing and Same-day Initiation of PrEP
Brief Title: Express Testing and Same-day Initiation of PrEP Study
Acronym: Express-PrEP
Status: Active, not recruiting | Type: Observational
Sponsor: HQ Toronto (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IN-CA-412-6433
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: HIV Prevention
Keywords: PrEP; HIV
MeSH Terms: interventions — emtricitabine tenofovir alafenamide; Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- gbMSM: This study will enroll gay, bisexual men who have sex with men (gbMSM), transgender and gender non-binary participants.
  Interventions: Drug: Descovy

INTERVENTIONS:
Drug: Descovy — Descovy is a once-daily prescription medicine for adults and adolescents at risk of HIV. It helps lower the chances of getting HIV through sex. In this study, patients at risk of acquiring HIV will be screened for HIV and those that are HIV-negative will be initiated on PrEP within 24 hours.
  Other Names: emtricitabine 200 mg/tenofovir alafenamide 25 mg

SUMMARY:
This study is an observational cohort study to measure the impact of express testing and same-day initiation of Pre-Exposure Prophylaxis (PrEP) on outcomes related to the PrEP cascade. The investigators expect that same day initiation for PrEP will improve PrEP uptake. The investigators hypothesize that baseline HIV test positivity will be higher than that of general testing for gbMSM in Ontario. This is a key indicator to determine whether this targeted approach is able to access the highest risk population.

DETAILED DESCRIPTION:
Gay, bisexual men who have sex with men (gbMSM) account for over half of new HIV infections in Canada each year, experience a disproportionately high burden of new HIV infections, and a 131-fold higher risk of HIV than other Canadian men. Transgender women (TGW) are a population also at increased HIV risk and a priority for HIV prevention.

Pre-Exposure Prophylaxis (PrEP) for prevention of HIV infection using regular oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) or tenofovir alafenamide/emtricitabine (TAF/FTC) is an effective and safe HIV prevention option for MSM and data from the Canadian setting shows that awareness, interest and willingness to use PrEP have been rising in this population. Accessing PrEP is currently a multistep process, often across several healthcare settings, that creates unnecessary barriers leading to attrition or delays in initiation. Although PrEP uptake has increased over time in Ontario, there is a significant proportion of gbMSM who are not on PrEP that would benefit from initiation. In multiple studies of the PrEP cascade, drop off in patient participation can be seen at each -level of the continuum often as a result of delays in the accessibility of starting PrEP and the multiple steps required by patients.

The success of PrEP has led to a decrease in HIV diagnoses among men in Ontario in recent years, however, Black and Latinx gbMSM, and TGW make up a disproportionate percentage of positive diagnoses. Despite recent increases in PrEP uptake, it is well understood that BIPOC experience barriers when accessing PrEP, leading to lower rates of uptake compared to white gbMSM. A critical component of the HIV care continuum in Ontario will be to increase the uptake of testing and PrEP use within those populations experiencing disproportionate risk, as well as people who experience mental health or substance use issues.

Currently in Ontario, the turnaround time between sample collection and a confirmatory positive HIV test to the provider can be a week or more. The HQ lab is designed to conduct laboratory HIV screening within 1 to 2 hours and confirmatory testing onsite in approximately 3 to 4 hours. This will allow the HQ team to offer same-day PrEP initiation for eligible participants in less than 2 hours following a negative HIV screening test. No other clinical program has been able to draw the blood sample, have both the screening and confirmatory lab-based testing done, give the diagnosis, and initiate PrEP on the same day.

ELIGIBILITY:
Inclusion Criteria:

Patients 16 years of age and older, visiting HQ for express testing, HIV negative and not currently on PrEP.

Exclusion criteria: Patients under the age of 16 years of age, currently on PrEP, or living with HIV.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is targeting gay, bisexual men who have sex with men, transgender, and gender non-binary individuals
Sampling Method: Non-Probability Sample
Enrollment: 816 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of PrEP in a rapid, same day treatment initiation setting. | January 2023 to January 2024
  The primary objective is to assess PrEP uptake in a rapid, same day treatment initiation setting. This includes proportion of those eligible for PrEP that initiate treatment on the same day as testing. All persons will be offered express laboratory testing onsite, which will greatly improve the time for PrEP initiation. Those people who test negative for HIV, and are eligible for PrEP based on a risk score, will be offered PrEP same day. The investigators expect that same day initiation for PrEP will improve PrEP uptake.

SECONDARY OUTCOMES:
Uptake of PrEP among key groups | January 2023 to January 2024
  The secondary objective is to measure PrEP uptake among key risk groups. HQ provides target testing programs for high risk people, including Black and Latinx gbMSM, transgender and gender non-binary individuals, as well as those who experience mental health concerns and use substances. The study will assess if same-day initiation for key groups will prevent loss to follow up and will enable higher PrEP uptake among stigmatized and marginalized communities.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Woodward, MD, Principal Investigator — HQ Health HubToronto
Locations (1):
- HQ Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There are not any current plans to share individual patient data with researchers in other institutions. If this were to take place, the data would be fully anonymized and proper data sharing agreements would be put in place.